CLINICAL TRIAL: NCT04127045
Title: ProspEctive Cohort Study on Integrated and Multidisciplinary Approach to Femur FRactures' manAgement in Over 65 Population
Brief Title: ProspEctive Cohort Study on Multidisciplinary Approach to Femur FRactures' manAgement in Over 65 Population
Acronym: EFFRA-65
Status: Completed | Type: Observational
Sponsor: Biagio Moretti, MD (Other)
Responsible Party: Sponsor-Investigator, Biagio Moretti, MD, Full Professor, University of Bari
Organization: University of Bari (Other)
Other Study IDs: 5559
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Hip Fractures; Intertrochanteric Fractures; Femur Fracture
Keywords: gait analysis; hip fracture; elderly; mobility
MeSH Terms: conditions — Hip Fractures; Femoral Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IMN-Group: Patients treated with intramedullary nailing
  Interventions: Procedure: IMN-Group
- HA-Group: Patients treated with Hemiarthroplasty
  Interventions: Procedure: HA-Group

INTERVENTIONS:
Procedure: IMN-Group — Most intertrochanteric fractures are managed with an intramedullary nail, which allows for impaction at the fracture site. The intramedullary nail is placed directly into the marrow canal of the bone through an opening made at the top of the greater trochanter. A lag screw is then placed through the nail and up into the neck and head of the hip. As with the compression hip screw, sliding of the lag screw and impaction of the fracture take place.
  Groups: IMN-Group
Procedure: HA-Group — In the older patient, the chance that the head of the femur is damaged in this way is higher. It is generally felt that for these displaced fractures, patients will do better if some of the components of the hip are replaced. In some cases, this can mean a replacement of the ball, or head of the femur (hemiarthroplasty).
  Groups: HA-Group

SUMMARY:
Hip fractures are an increasing public health concern as the population continues to age. The increased morbidity and mortality in the 12-month period after hip fracture is largely related to decreased mobility. However, very few studies have analyzed the radiographic factors associated with gait impairment after intertrochanteric hip fractures. This study evaluates gait and mobility after surgical fixation of IT fractures in elderly population with Gait Analysis in combination with clinical and radiographic information.

DETAILED DESCRIPTION:
Hip fractures are an increasing public health concern as the population continues to age. The increased morbidity and mortality in the 12-month period after hip fracture is largely related to decreased mobility. However, very few studies have analyzed the radiographic factors associated with gait impairment after InterTrochanteric (IT) hip fractures. Improving gait and mobility after surgical fixation of IT fractures is one important target of research efforts.

All the patients with IT hip fractures (AO/OTA 31) treated between October 2017 and April 2018 were enrolled. Inclusion criteria consisted of age older than 65 years, previous walking ability, no neurological disease and no other musculoskeletal disorders. The study was approved by the institutional review board of the Local Ethical Committee (reference number 5559). All patients provided written informed consent for participation in the study.

All patients were treated with intramedullary nailing (IMN) or hemiarthroplasty (HA) according to the current international guidelines and to their clinical history.

Radiographs were analyzed at the time of surgery and at each follow-up visit. Clinical outcomes were assessed according to the Harris Hip Score (HHS) and Western Ontario and Mc Master University (WOMAC).

At 6- and 12-months follow-up appointments, gait parameters were measured and recorded in our Gait Analysis Laboratory (BTS Bioengineering SpA, Italy) located in AOUC Policlinico di Bari (Rehabilitation Unit). All participants performed several walking trials at their natural speed. All patients were fitted with full-body external reflective markers placed according to Davis' procedures. A static video trial was recorded with subjects positioned in a neutral standing posture to create a reference for defining neutral joint angles.

In addition, at 12-months follow-up, dual energy X-ray absorptiometry (DXA) has been acquired in order to collect T-score data.

Statistical analyses were performed using IBM SPSS version 23. A p value of <0.05 was considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* age older than 65 years
* previous walking ability
* surgical procedure (intramedullary nailing or hemiarthroplasty)

Exclusion Criteria:

* neurological diseases
* musculoskeletal disorders
* cardiovascular diseases

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: All the patients with IT hip fractures (AO/OTA 31) treated between October 2017 and April 2018 in the Orthopedic and Trauma Unit of AOUC Policlinico di Bari were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in HHS at follow-up | 12- months
  Harris Hip Score gives a maximum of 100 points. Pain receives 44 points, function 47 points, range of motion 5 points, and deformity 4 points. Function is subdivided into activities of daily living (14 points) and gait (33 points). The higher the HHS, the less dysfunction.
Changes in WOMAC at follow-up | 12- months
  Western Ontario and Mc Master University Scale evaluates the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints. The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. The higher the score, the poorer the function. Therefore, an improvement was achieved by reducing the overall score.
Changes in T-Score at follow-up | 12- months
  T-score is the relevant measure when screening for osteoporosis extracted from Dual energy X-ray Absorptiometry (DXA). It is the bone mineral density (BMD) at the site when compared to the young normal reference mean. A T-score between +1 and -1 is considered normal or healthy. A T-score between -1 and -2.5 indicates that you have low bone mass, although not low enough to be diagnosed with osteoporosis. A T-score of -2.5 or lower indicates that you have osteoporosis. The greater the negative number, the more severe the osteoporosis.
Changes in Spatial Parameters of Gait at follow-up | 12- months
  Gait Analysis will be performed in two different time points and parameters related to spatial characteristics of gait during a gait cycle will be estimated: stride length (m), step length (m), step width (m).
Changes in Temporal Parameters of Gait at follow-up | 12- months
  Gait Analysis will be performed in two different time points and parameters related to temporal characteristics of gait during a gait cycle will be estimated (expressed in percentage): stance phase (%), swing phase (%)

SECONDARY OUTCOMES:
Changes in ROM of Kinematic Angles | 12- months
  Gait Analysis will be performed in two different time points and the changes in ankle, knee, hip and pelvis angles (all measured in degree) will be estimated.
GGA-g Index | 12- months
  Gait Analysis will be performed in two different time points and an overall index of asymmetry (Global Gait Asymmetry) during the gait cycle will be estimated. The higher the index, the higher the asymmetry between body part.
GGA-a Index | 12- months
  Gait Analysis will be performed in two different time points and an index of asymmetry (Global Gait Asymmetry) during the gait cycle in each kinematic angles (ankle, knee, hip and pelvis) will be estimated. The higher the index, the higher the asymmetry between body part.

CONTACTS AND LOCATIONS:
Overall Officials: Biagio Moretti, M.D., Principal Investigator — University of Bari
Locations (1):
- Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari, Bari, IT, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bortone, I., Caringella, N., Lelli, G., Rifino, F., Di Candia, A., Fiore, P., & Moretti, B. (2018). Effective mobility recovery after femoral neck fractures: The necessity of gait analysis in the immediate post-operative aftercare. Gait & Posture, 66, S7.
- [Result] Bizzoca D, Bortone I, Vicenti G, Caringella N, Rifino F, Moretti B. Gait analysis in the postoperative assessment of intertrochanteric femur fractures. J Biol Regul Homeost Agents. 2020 Jul-Aug;34(4 Suppl. 3):345-351. Congress of the Italian Orthopaedic Research Society. PMID 33261299